CLINICAL TRIAL: NCT05346445
Title: Citalopram Improves Vasomotor and Urogenital Syndromes in Mexican Patients With Post-menopause
Brief Title: Comparison of Fluoxetine Versus Citalopram Therapy to Control Postmenopausal Vasomotor Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Regional 1o de Octubre (Other)
Collaborators: Universidad Nacional Autonoma de Mexico (Other); National Polytechnic Institute, Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 122.2021
Record Dates: First submitted 2022-04-14; First posted 2022-04-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Postmenopause; Hot Flashes
Keywords: Postmenopause; Fluoxetine; Menopause Rating Scale; Vasomotor syndrome; Urogenital syndrome; Citalopram; Non hormonal therapy; Non-hormonal therapies; Serotonin reuptake inhibitors
MeSH Terms: conditions — Hot Flashes | interventions — Fluoxetine; Citalopram

STUDY DESIGN:
Intervention Model Description: This study was a prospective randomized clinical trial made in Mexican women diagnosed with postmenopause from the climacteric clinic of the regional hospital "1ro de Octubre-Instituto de Seguridad y Servicios Sociales para los Trabajadores del Estado (ISSSTE)". Eligible participants were randomly selected in each consult to receive citalopram 20 mg/d or fluoxetine 20 mg/d for six months. The evaluation of the MRS score was done at the first consult and three and six months after medication. The institutional ethical committee of the hospital approved the study on May 20th, 2021, with registration number CONBIOETICA-09-CEI-012-20170421 and the internal registration number 122.2021. All participants provided written informed consent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluoxetine group (Active Comparator): Participants received fluoxetine, 20 mg tablets, once a day for six months.
  Interventions: Drug: Fluoxetine 20 MG
- Citalopram group (Experimental): Participants received citalopram, 20 mg tablets, once a day for six months.
  Interventions: Drug: Citalopram 20mg

INTERVENTIONS:
Drug: Fluoxetine 20 MG — Participants received non-hormonal treatment with fluoxetine.
  Other Names: Generic PISA®
  Arms: Fluoxetine group
Drug: Citalopram 20mg — Participants received non-hormonal treatment with citalopram.
  Other Names: PREPRAM®
  Arms: Citalopram group

SUMMARY:
This study determined the efficacy of non-hormonal therapy with citalopram compared to fluoxetine, for the treatment of menopausal symptoms in Mexican women with vasomotor syndrome (VMS) and urogenital syndrome.

DETAILED DESCRIPTION:
Women's reproductive life goes through a senescence process called transition to menopause, which generates an imbalance in estrogenic hormonal regulation that is more evident between the fifth and sixth decades of life. This condition allows the passage from an active reproductive stage to an inactive one, which triggers an adaptative physiological response to the reduction of estrogens. However, the progressive depletion of estrogen levels causes clinical signs and symptoms in the central nervous system, metabolism, musculoskeletal apparatus, urogenital system, and skin. These symptoms lead to disability, work absenteeism, and health costs, affecting the quality of life of women in this stage. Vasomotor symptoms are the main clinical manifestation for which women seek treatment. Vasomotor syndrome (VMS) occurs in 75 to 80% of all women. The first-line management of menopausal symptoms is hormone replacement therapy (HRT). However, some patients present adverse effects or contraindications for using it.

The aim of this study was to determine the efficacy of the citalopram for treating menopausal symptoms in Mexican women with vasomotor syndrome (VMS) and urogenital syndrome.

This study was a prospective randomized clinical trial, where 91 post-menopausal participants with severe baseline scores on the Menopause Rating Scale (MRS) were randomly selected and treated with citalopram (n=49) or fluoxetine (n=42). Changes from baseline MRS score at three and six months of treatment were evaluated.

Participants were randomly assigned to groups before each consult. Randomization was done using RAND and RANK functions from Excel-Word to generate unique random numbers for every participant´s ID. Fluoxetine is the Gold Standard treatment in Mexico, whereby it was used as the control medication. Loading doses of citalopram 20 mg orally or fluoxetine 20 mg orally were administrated.

Statical analysis was performed using PAST 3.0 and GraphPad Prism 8.4.3. software. Some statical parameters, such as arithmetic median (µ), standard deviation (S.D.), and Hazard ratio, were calculated using Excel-Word. Graphics were constructed with GraphPad Prism 8.4.3. Tables and Forest plots were done in Excel-Word. Odds ratio (OR), Relative Risk (RR), and chi-squared were calculated with PAST 3.0 software. The assigned α value for this study was <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Participants who attended the climacteric consultation for the first time, without prior treatment of menopausal symptoms, and who met postmenopausal criteria.
* Participants who met the criteria for vasomotor syndrome and score greater than 17 points in total MRS.
* Participants without psychiatric pathology (psychiatric illnesses such as major depression, generalized anxiety disorder, among others).
* Participants who agreed to participate and gave their written informed consent.

Exclusion Criteria:

* Participants who had contraindications to receive serotonin reuptake inhibitors (SSRIs).
* Participants who were receiving prior treatment for the postmenopausal or vasomotor syndrome.
* Participants who did not agree to participate or sign the informed consent.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline Menopause Rating Scale (MRS) total score at 3 months | 3 months
  Menopause Rating Scale measures the severity of ageing symptoms and their impact on Health-Related Quality of Life. It considers the score of the somatic, urogenital, and psychological domains. A score of 0-4 was considered minimal severity, 5-8 mild, 9-16 moderate, and greater than 17 severe.
Change from baseline Menopause Rating Scale (MRS) total score at 6 months | 6 months
  Menopause Rating Scale measures the severity of ageing symptoms and their impact on Health-Related Quality of Life. It considers the score of the somatic, urogenital, and psychological domains. A score of 0-4 was considered minimal severity, 5-8 mild, 9-16 moderate, and greater than 17 severe.
Change from baseline Menopause Rating Scale (MRS) somatic domain score at 3 months | 3 months
  It considers the score obtained from the somatic dimension, which includes hot flashes, heart problems, sleep problems, and muscle and joint pain. A score of 0-2 was considered minimal severity, 3-4 mild, 5-8 moderate, and greater than 9 severe.
Change from baseline Menopause Rating Scale (MRS) somatic domain score at 6 months | 6 months
  It considers the score obtained from the somatic dimension, which includes hot flashes, heart problems, sleep problems, and muscle and joint pain. A score of 0-2 was considered minimal severity, 3-4 mild, 5-8 moderate, and greater than 9 severe.
Change from baseline Menopause Rating Scale (MRS) urogenital domain score at 3 months | 3 months
  It considers the score obtained from the urogenital dimension, which includes sexual problems, bladder problems and vaginal dryness. A score of 0 was considered minimal severity, 1 mild, 2-3 moderate, and greater than 4 severe.
Change from baseline Menopause Rating Scale (MRS) urogenital domain score at 6 months | 6 months
  It considers the score obtained from the urogenital dimension, which includes sexual problems, bladder problems and vaginal dryness. A score of 0 was considered minimal severity, 1 mild, 2-3 moderate, and greater than 4 severe.
Change from baseline Menopause Rating Scale (MRS) psychological domain score at 3 months | 3 months
  It considers the score obtained from the psychological dimension, which includes depression, irritability, anxiety and tiredness. A score of 0-1 was considered minimal severity, 2-3 mild, 4-6 moderate, and greater than 7 severe.
Change from baseline Menopause Rating Scale (MRS) psychological domain score at 6 months | 6 months
  It considers the score obtained from the psychological dimension, which includes depression, irritability, anxiety and tiredness. A score of 0-1 was considered minimal severity, 2-3 mild, 4-6 moderate, and greater than 7 severe.
Change from baseline score in Item 1 of the Menopause Rating Scale (MRS) at 3 months | 3 months
  Item 1 considers the score obtained from hot flashes on the MRS scale. 0 points were assigned if the participants reported no symptoms, 1 point if they reported mild symptoms, 2 points if they reported moderate symptoms, 3 points if they reported severe symptoms, and 4 points if they reported extremely severe symptoms.
Change from baseline score in Item 1 of the Menopause Rating Scale (MRS) at 6 months | 3 months
  Item 1 considers the score obtained from hot flashes on the MRS scale. 0 points were assigned if the participants reported no symptoms, 1 point if they reported mild symptoms, 2 points if they reported moderate symptoms, 3 points if they reported severe symptoms, and 4 points if they reported extremely severe symptoms.

SECONDARY OUTCOMES:
Change from the severity of individual Menopause Rating Scale (MRS) items at 6 months | 6 months
  It considers the obtained score from individual MRS items. 0 points were assigned if the participants reported no symptoms, 1 point if they reported mild symptoms, 2 points if they reported moderate symptoms, 3 points if they reported severe symptoms, and 4 points if they reported extremely severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Ocampo-Godinez, M.D., Ph.D., Study Director — Tissue Bioengineering Laboratory, National Autonomous University of Mexico [UNAM]; Patricia Loranca-Moreno, M.D., M.Sc., Study Director — Peri-postmenopause and bone metabolism clinic. Regional Hospital October 1st ISSSTE; Alan Rios-Espinosa, M.D., Principal Investigator — Peri-postmenopause and bone metabolism clinic. Regional Hospital October 1st ISSSTE
Locations (1):
- Peri-postmenopause and bone metabolism clinic. Regional Hospital October 1st ISSSTE, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El Khoudary SR, McClure CK, VoPham T, Karvonen-Gutierrez CA, Sternfeld B, Cauley JA, Khalil N, Sutton-Tyrrell K. Longitudinal assessment of the menopausal transition, endogenous sex hormones, and perception of physical functioning: the Study of Women's Health Across the Nation. J Gerontol A Biol Sci Med Sci. 2014 Aug;69(8):1011-7. doi: 10.1093/gerona/glt285. Epub 2014 Jan 24. PMID 24465026
- [Background] Jones CM, Boelaert K. The Endocrinology of Ageing: A Mini-Review. Gerontology. 2015;61(4):291-300. doi: 10.1159/000367692. Epub 2014 Nov 27. PMID 25471682
- [Background] Blumel JE, Lavin P, Vallejo MS, Sarra S. Menopause or climacteric, just a semantic discussion or has it clinical implications? Climacteric. 2014 Jun;17(3):235-41. doi: 10.3109/13697137.2013.838948. Epub 2013 Nov 7. PMID 23998690
- [Background] Monteleone P, Mascagni G, Giannini A, Genazzani AR, Simoncini T. Symptoms of menopause - global prevalence, physiology and implications. Nat Rev Endocrinol. 2018 Apr;14(4):199-215. doi: 10.1038/nrendo.2017.180. Epub 2018 Feb 2. PMID 29393299
- [Background] Kim MJ, Yim G, Park HY. Vasomotor and physical menopausal symptoms are associated with sleep quality. PLoS One. 2018 Feb 20;13(2):e0192934. doi: 10.1371/journal.pone.0192934. eCollection 2018. PMID 29462162
- [Background] Sarrel P, Portman D, Lefebvre P, Lafeuille MH, Grittner AM, Fortier J, Gravel J, Duh MS, Aupperle PM. Incremental direct and indirect costs of untreated vasomotor symptoms. Menopause. 2015 Mar;22(3):260-6. doi: 10.1097/GME.0000000000000320. PMID 25714236
- [Background] Avis NE, Crawford SL, Green R. Vasomotor Symptoms Across the Menopause Transition: Differences Among Women. Obstet Gynecol Clin North Am. 2018 Dec;45(4):629-640. doi: 10.1016/j.ogc.2018.07.005. Epub 2018 Oct 25. PMID 30401547
- [Background] Langer RD, Hodis HN, Lobo RA, Allison MA. Hormone replacement therapy - where are we now? Climacteric. 2021 Feb;24(1):3-10. doi: 10.1080/13697137.2020.1851183. Epub 2021 Jan 6. PMID 33403881
- [Background] Deecher DC, Dorries K. Understanding the pathophysiology of vasomotor symptoms (hot flushes and night sweats) that occur in perimenopause, menopause, and postmenopause life stages. Arch Womens Ment Health. 2007;10(6):247-57. doi: 10.1007/s00737-007-0209-5. Epub 2007 Dec 12. PMID 18074100
- [Background] De Franciscis P, Cobellis L, Fornaro F, Sepe E, Torella M, Colacurci N. Low-dose hormone therapy in the perimenopause. Int J Gynaecol Obstet. 2007 Aug;98(2):138-42. doi: 10.1016/j.ijgo.2007.04.008. Epub 2007 Jun 18. PMID 17572422
- [Background] Stubbs C, Mattingly L, Crawford SA, Wickersham EA, Brockhaus JL, McCarthy LH. Do SSRIs and SNRIs reduce the frequency and/or severity of hot flashes in menopausal women. J Okla State Med Assoc. 2017 May;110(5):272-274. PMID 28649145
- [Background] Kapoor E, Faubion S, Hurt RT, Fischer K, Schroeder D, Fokken S, Croghan IT. A selective serotonin receptor agonist for weight loss and management of menopausal vasomotor symptoms in overweight midlife women: a pilot study. Menopause. 2020 Nov;27(11):1228-1235. doi: 10.1097/GME.0000000000001599. PMID 33110038
- [Background] Ensrud KE, Joffe H, Guthrie KA, Larson JC, Reed SD, Newton KM, Sternfeld B, Lacroix AZ, Landis CA, Woods NF, Freeman EW. Effect of escitalopram on insomnia symptoms and subjective sleep quality in healthy perimenopausal and postmenopausal women with hot flashes: a randomized controlled trial. Menopause. 2012 Aug;19(8):848-55. doi: 10.1097/gme.0b013e3182476099. PMID 22433978
- [Background] Wroolie TE, Williams KE, Keller J, Zappert LN, Shelton SD, Kenna HA, Reynolds MF, Rasgon NL. Mood and neuropsychological changes in women with midlife depression treated with escitalopram. J Clin Psychopharmacol. 2006 Aug;26(4):361-6. doi: 10.1097/01.jcp.0000227699.26375.f8. PMID 16855452
- [Background] Shams T, Firwana B, Habib F, Alshahrani A, Alnouh B, Murad MH, Ferwana M. SSRIs for hot flashes: a systematic review and meta-analysis of randomized trials. J Gen Intern Med. 2014 Jan;29(1):204-13. doi: 10.1007/s11606-013-2535-9. Epub 2013 Jul 26. PMID 23888328
- [Background] Soares CN, Arsenio H, Joffe H, Bankier B, Cassano P, Petrillo LF, Cohen LS. Escitalopram versus ethinyl estradiol and norethindrone acetate for symptomatic peri- and postmenopausal women: impact on depression, vasomotor symptoms, sleep, and quality of life. Menopause. 2006 Sep-Oct;13(5):780-6. doi: 10.1097/01.gme.0000240633.46300.fa. PMID 16894334
- [Background] Suvanto-Luukkonen E, Koivunen R, Sundstrom H, Bloigu R, Karjalainen E, Haiva-Mallinen L, Tapanainen JS. Citalopram and fluoxetine in the treatment of postmenopausal symptoms: a prospective, randomized, 9-month, placebo-controlled, double-blind study. Menopause. 2005 Jan-Feb;12(1):18-26. doi: 10.1097/00042192-200512010-00006. PMID 15668596
- [Background] Barton DL, LaVasseur BI, Sloan JA, Stawis AN, Flynn KA, Dyar M, Johnson DB, Atherton PJ, Diekmann B, Loprinzi CL. Phase III, placebo-controlled trial of three doses of citalopram for the treatment of hot flashes: NCCTG trial N05C9. J Clin Oncol. 2010 Jul 10;28(20):3278-83. doi: 10.1200/JCO.2009.26.6379. Epub 2010 May 24. PMID 20498389
- [Background] Soares CN, Poitras JR, Prouty J, Alexander AB, Shifren JL, Cohen LS. Efficacy of citalopram as a monotherapy or as an adjunctive treatment to estrogen therapy for perimenopausal and postmenopausal women with depression and vasomotor symptoms. J Clin Psychiatry. 2003 Apr;64(4):473-9. doi: 10.4088/jcp.v64n0419. PMID 12716252
- [Background] Rathnayake N, Lenora J, Alwis G, Lekamwasam S. Cross cultural adaptation and analysis of psychometric properties of Sinhala version of Menopause Rating Scale. Health Qual Life Outcomes. 2018 Aug 6;16(1):161. doi: 10.1186/s12955-018-0977-9. PMID 30081962
- [Background] Jahangiry L, Parviz R, Mirghafourvand M, Khazaee-Pool M, Ponnet K. The psychometric properties of the Persian menopause rating scale. BMC Womens Health. 2020 Aug 12;20(1):172. doi: 10.1186/s12905-020-01027-0. PMID 32787824
- [Background] Ajani K, Nimavat D, Vidja M, Moradiya A, Panchasara D, Bhalodiya S, Miyatra K, Tank KD. Translation, Reliability, and Validity Test of Gujarati Version of Menopause Rating Scale in Postmenopausal Women for Menopause-Related Symptoms. Indian J Community Med. 2021 Jan-Mar;46(1):40-44. doi: 10.4103/ijcm.IJCM_163_20. Epub 2021 Mar 1. PMID 34035574
- [Background] Anagnostis P, Bitzer J, Cano A, Ceausu I, Chedraui P, Durmusoglu F, Erkkola R, Goulis DG, Hirschberg AL, Kiesel L, Lopes P, Pines A, van Trotsenburg M, Lambrinoudaki I, Rees M. Menopause symptom management in women with dyslipidemias: An EMAS clinical guide. Maturitas. 2020 May;135:82-88. doi: 10.1016/j.maturitas.2020.03.007. Epub 2020 Mar 16. PMID 32209279
- [Background] Guthrie KA, Larson JC, Ensrud KE, Anderson GL, Carpenter JS, Freeman EW, Joffe H, LaCroix AZ, Manson JE, Morin CM, Newton KM, Otte J, Reed SD, McCurry SM. Effects of Pharmacologic and Nonpharmacologic Interventions on Insomnia Symptoms and Self-reported Sleep Quality in Women With Hot Flashes: A Pooled Analysis of Individual Participant Data From Four MsFLASH Trials. Sleep. 2018 Jan 1;41(1):zsx190. doi: 10.1093/sleep/zsx190. PMID 29165623
- [Background] Belso N, Kiss K, Rihmer Z, Tuzko N, Toth SJ, Paulin F. Major depressive disorder and response to citalopram treatment in women attending menopause clinic. Int J Psychiatry Clin Pract. 2003;7(4):269-72. doi: 10.1080/13651500310003183. PMID 24930413
- [Background] Freeman MP, Hill R, Brumbach BH. Escitalopram for perimenopausal depression: an open-label pilot study. J Womens Health (Larchmt). 2006 Sep;15(7):857-61. doi: 10.1089/jwh.2006.15.857. PMID 16999641
- [Background] Soares CN, Thase ME, Clayton A, Guico-Pabia CJ, Focht K, Jiang Q, Kornstein SG, Ninan P, Kane CP, Cohen LS. Desvenlafaxine and escitalopram for the treatment of postmenopausal women with major depressive disorder. Menopause. 2010 Jul;17(4):700-11. doi: 10.1097/gme.0b013e3181d88962. PMID 20539246
- [Background] Barton DL, Loprinzi CL, Novotny P, Shanafelt T, Sloan J, Wahner-Roedler D, Rummans TA, Christensen B, Dakhill SR, Martin LS. Pilot evaluation of citalopram for the relief of hot flashes. J Support Oncol. 2003 May-Jun;1(1):47-51. PMID 15352642
- [Background] Defronzo Dobkin R, Menza M, Allen LA, Marin H, Bienfait KL, Tiu J, Howarth J. Escitalopram reduces hot flashes in nondepressed menopausal women: A pilot study. Ann Clin Psychiatry. 2009 Apr-Jun;21(2):70-6. PMID 19439155
- [Background] Freedman RR, Kruger ML, Tancer ME. Escitalopram treatment of menopausal hot flashes. Menopause. 2011 Aug;18(8):893-6. doi: 10.1097/gme.0b013e31820ccae9. PMID 21540755
- [Background] LaCroix AZ, Freeman EW, Larson J, Carpenter JS, Joffe H, Reed SD, Newton KM, Seguin RA, Sternfeld B, Cohen L, Ensrud KE. Effects of escitalopram on menopause-specific quality of life and pain in healthy menopausal women with hot flashes: a randomized controlled trial. Maturitas. 2012 Dec;73(4):361-8. doi: 10.1016/j.maturitas.2012.09.006. Epub 2012 Sep 30. PMID 23031421
- [Background] Carpenter JS, Guthrie KA, Larson JC, Freeman EW, Joffe H, Reed SD, Ensrud KE, LaCroix AZ. Effect of escitalopram on hot flash interference: a randomized, controlled trial. Fertil Steril. 2012 Jun;97(6):1399-404.e1. doi: 10.1016/j.fertnstert.2012.03.001. Epub 2012 Apr 3. PMID 22480818
- [Background] Joffe H, Guthrie KA, Larson J, Cohen LS, Carpenter JS, Lacroix AZ, Freeman EW. Relapse of vasomotor symptoms after discontinuation of the selective serotonin reuptake inhibitor escitalopram: results from the menopause strategies: finding lasting answers for symptoms and health research network. Menopause. 2013 Mar;20(3):261-8. doi: 10.1097/GME.0b013e31826d3108. PMID 23435022
- [Background] Diem SJ, LaCroix AZ, Reed SD, Larson JC, Newton KM, Ensrud KE, Woods NF, Guthrie KA. Effects of pharmacologic and nonpharmacologic interventions on menopause-related quality of life: a pooled analysis of individual participant data from four MsFLASH trials. Menopause. 2020 Oct;27(10):1126-1136. doi: 10.1097/GME.0000000000001597. PMID 32701665
- [Background] Freeman EW, Guthrie KA, Caan B, Sternfeld B, Cohen LS, Joffe H, Carpenter JS, Anderson GL, Larson JC, Ensrud KE, Reed SD, Newton KM, Sherman S, Sammel MD, LaCroix AZ. Efficacy of escitalopram for hot flashes in healthy menopausal women: a randomized controlled trial. JAMA. 2011 Jan 19;305(3):267-74. doi: 10.1001/jama.2010.2016. PMID 21245182
- [Background] Davari-Tanha F, Soleymani-Farsani M, Asadi M, Shariat M, Shirazi M, Hadizadeh H. Comparison of citalopram and venlafaxine's role in treating sleep disturbances in menopausal women, a randomized, double-blind, placebo-controlled trial. Arch Gynecol Obstet. 2016 May;293(5):1007-13. doi: 10.1007/s00404-015-3900-1. Epub 2015 Oct 5. PMID 26437957
- [Background] Shirazi M, Jalalian MN, Abed M, Ghaemi M. The Effectiveness of Melissa Officinalis L. versus Citalopram on Quality of Life of Menopausal Women with Sleep Disorder: A Randomized Double-Blind Clinical Trial. Rev Bras Ginecol Obstet. 2021 Feb;43(2):126-130. doi: 10.1055/s-0040-1721857. Epub 2021 Jan 19. PMID 33465795
- [Background] Molaie M, Darvishi B, Jafari Azar Z, Shirazi M, Amin G, Afshar S. Effects of a combination of Nigella sativa and Vitex agnus-castus with citalopram on healthy menopausal women with hot flashes: results from a subpopulation analysis. Gynecol Endocrinol. 2019 Jan;35(1):58-61. doi: 10.1080/09513590.2018.1499086. Epub 2018 Aug 21. PMID 30129806
- [Background] Valdes-Sustaita B, Lopez-Rubalcava C, Gonzalez-Trujano ME, Garcia-Viguera C, Estrada-Camarena E. Aqueous Extract of Pomegranate Alone or in Combination with Citalopram Produces Antidepressant-Like Effects in an Animal Model of Menopause: Participation of Estrogen Receptors. Int J Mol Sci. 2017 Dec 19;18(12):2643. doi: 10.3390/ijms18122643. PMID 29257042
- [Background] Zhou J, Wang X, Feng L, Xiao L, Yang R, Zhu X, Shi H, Hu Y, Chen R, Boyce P, Wang G. Venlafaxine vs. fluoxetine in postmenopausal women with major depressive disorder: an 8-week, randomized, single-blind, active-controlled study. BMC Psychiatry. 2021 May 19;21(1):260. doi: 10.1186/s12888-021-03253-8. PMID 34011310
- [Derived] Rios-Espinosa A, Cruz-Luna M, Garmendia-Gallardo C, Hernandez-Castanon MY, Hernandez-Hernandez VY, Sanchez-Tinoco PM, Bajonero-Dominguez A, Vergara Lope-Nunez JA, Alvarez-Perez MA, Gonzalez-Quiroz JL, Loranca-Moreno P, Ocampo-Godinez JM. Citalopram improves vasomotor syndrome and urogenital syndrome of menopause in Mexican women: a randomized clinical trial. Arch Gynecol Obstet. 2022 Dec;306(6):2035-2045. doi: 10.1007/s00404-022-06732-9. Epub 2022 Aug 23. PMID 35997971